CLINICAL TRIAL: NCT01256554
Title: Phase I Study of Feasibility of Single Session Spine Stereotactic Radiosurgery (SSRS) in the Primary Management of Patients With Inoperable, Previously Irradiated Metastatic Epidural Spinal Cord Compression (MESCC)
Brief Title: Single Session Spine Stereotactic Radiosurgery in Metastatic Epidural Spinal Cord Compression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0653; NCI-2011-00273 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Epidural Spinal Cord Compression
Keywords: Stereotactic Radiosurgery; SSRS; Radiation; Radiotherapy; Metastatic Epidural Spinal Cord Compression; MESCC
MeSH Terms: interventions — Radiosurgery; Radiation; Radiotherapy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Radiosurgery (SSRS) (Experimental): Target dose of 18 or 24 Gy to spine in single session of radiation. Questionnaire completion about health symptoms and pain at baseline, 3 months, 6 months, 9 months, 12 months, 24 months, then every 6 months.
  Interventions: Procedure: Stereotactic Radiosurgery (SSRS); Behavioral: Questionnaires

INTERVENTIONS:
Procedure: Stereotactic Radiosurgery (SSRS) — Target dose of 18 or 24 Gy to spine in single session of radiation.
  Other Names: Stereotactic Radiosurgery; SSRS; Radiation; Radiotherapy; Metastatic Epidural Spinal Cord Compression; MESCC
Behavioral: Questionnaires — Questionnaire completion about health symptoms and pain at baseline, 3 months, 6 months, 9 months, 12 months, 24 months, then every 6 months.
  Other Names: Surveys

SUMMARY:
The goal of this clinical study is to learn the feasibility of using a single session of radiation, known as spine stereotactic radiosurgery (SSRS), to treat metastatic epidural spinal cord compression.

DETAILED DESCRIPTION:
Spinal cord compression is often treated with surgery followed by radiation in small doses every day for a number of days. When a patient cannot or will not have surgery, radiation is given daily. With increased accuracy and precision, higher doses of radiation can be given in a single session. Giving a higher dose in a single session may increase the chance that the tumor will stop growing into the spinal canal and will prevent spinal cord injury. This study will also help to identify the tolerance of the spinal cord to radiation in a single session.

Spine Stereotactic Radiosurgery:

You will lie in the mold that was made for you for 45-120 minutes while you receive your radiation treatment.

Follow-up Visits:

You will have follow-up visits at Months 3 (+/-2 weeks ), 6 (+/-4 weeks), 9 (+/-4 weeks), 12 (+/-8 weeks), 18 (+/-8 weeks), and 24 (+/-8 weeks) and then every 6 months after that. At each follow-up visit:

* Your medical history will be recorded, including usage of steroids.
* You will have a neurological exam.
* You will complete the 3 questionnaires about health, symptoms you may be having, and about pain.
* You will have an MRI of the spine.

If you are unable to return for follow-up clinic visits, you will be called and asked about your medical history, and you will complete the 3 questionnaires about your health, symptoms you may be having, and about pain. This call should take about 20 minutes.

Length of Study:

Your treatment will last 1 day. You will continue having follow-up visits or phone calls for as long as possible.

This is an investigational study. SSRS is FDA approved. The use of SSRS to treat metastatic epidural spinal cord compression is investigational.

Up to 36 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years old
2. Radiographically documented metastatic epidural compression on spine Magnetic resonance imaging (MRI) within 4 weeks of registration, defined radiographically, ranging from minimal canal compromise and thecal indentation to actual displacement of the spinal cord.
3. Maximum of 3 contiguous vertebral levels involved with metastasis in the spine to be irradiated in a single session
4. Signed Informed consent for irradiation
5. Diagnosis of cancer including but not limited to non-small cell lung cancer, breast, prostate, renal cell, melanoma, gastrointestinal, sarcoma, thyroid, head and neck primary, and unknown primary tumors
6. Motor Strength >/= 4 out of 5 in extremity or extremities affected by the level of the spinal cord compression
7. Karnofsky performance status (KPS) >/= 40
8. Patients deemed to be inoperable due to patient refusal, by neurosurgical evaluation, or for any reason
9. 1 prior course of spine radiotherapy to the current region of interest

Exclusion Criteria:

1. Prior irradiation of the site to be treated </= 3 months prior to registration
2. Inability to tolerate lying flat on treatment table for greater than 30 minutes.
3. Patients unable to undergo MRI of the spine
4. Patients who have previously received maximum cord tolerance of 45 Gy in 5 weeks conventional fractionation or similar biologically effective dose (BED) to the area of the spine to be treated. Below are the normalized BED at 2 Gy per fraction with alpha/beta=2 for spinal cord in commonly used fractionation schemes in previously irradiated patients. Conventional Radiotherapy (Normalized Biologically Effective Dose) 20 Gy in 5 fractions(30 Gy 2/2), 30 Gy in 10 fractions(37.5 Gy 2/2), 37.5 Gy in 15 fractions(42 Gy 2/2), 40 Gy in 20 fractions(40 Gy 2/2), 45 Gy in 25 fractions(43 Gy 2/2), 50 Gy in 25 fractions(50 Gy 2/2) following equation: nBED is calculated by dividing BED by (1 + d/a/b), where d is 2 Gy and for spinal cord late effect a/b is 2, and we describe the units as Gy 2/2 (i.e., Gy 2/2 = 2-Gy equivalent with a/b = 2)
5. Patients who are pregnant.
6. Patients who have cord compression from bone components or configuration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-12-03 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Number of Occurrences of Paralysis Caused by Radiation Myelitis (RM) | Up to 12 months following radiation
  Maximum acceptable Dmax will be that in which there are fewer RM events than TP events prior to 12 months and less than 2 RM events.

CONTACTS AND LOCATIONS:
Overall Officials: Amol J. Ghia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org